CLINICAL TRIAL: NCT02323035
Title: Investigative Headgear With CPAP Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIA150
Record Dates: First submitted 2014-12-15; First posted 2014-12-23 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Extraoral Traction Appliances

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Headgear (Experimental): Investigative Headgear with CPAP Mask.
  Interventions: Device: Headgear

INTERVENTIONS:
Device: Headgear — Investigative Headgear with CPAP Mask.

SUMMARY:
This investigation is designed to evaluate the at-home usability, performance, user acceptance and reliability of the Headgear with a CPAP Mask for a duration of 2-4 weeks.

DETAILED DESCRIPTION:
Up to 300 participants will be recruited for the trial, consisting of male and female participants diagnosed with OSA and receiving CPAP or Bi-level PAP for the treatment of their OSA. These include current CPAP mask users.

ELIGIBILITY:
Inclusion Criteria:

* AHI≥5 from the diagnostic night
* ≥18 years of age
* Prescribed CPAP or Bilevel therapy for OSA
* Existing CPAP mask users

Exclusion Criteria:

* Inability to give informed consent
* Patient intolerant to PAP
* Anatomical or physiological conditions making PAP therapy inappropriate
* History of respiratory disease or CO2 retention.
* Pregnant or think they may be pregnant
* Investigated by Land Transport Safety Authority

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Participants perception of the headgear on mask performance | 2-4 weeks
  Assess if the headgear with mask changes the perception of the performance of the mask.

SECONDARY OUTCOMES:
Number of participants that choose this Headgear over their usual. | 2-4 weeks
  Assess the acceptability of the headgear with mask.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavi Ogra, BSc, Principal Investigator — Clinical Research Scientist
Locations (1):
- Fisher & Paykel Healthcare, Auckland, New Zealand